CLINICAL TRIAL: NCT05192902
Title: Pain Perception Following Computer-Controlled vs. Conventional Dental Anesthesia: Randomized Controlled Trial
Brief Title: Pain Perception Following Computer-Controlled vs. Conventional Dental Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Sameh Attia, Head of the Dental Polyclinic, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCLA
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Pain Perception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Student-administered (Experimental)
  Interventions: Device: Computer-controlled Local Anaesthesia (CCLA); Device: Conventional Local Anaesthesia
- Dentist-administered (Placebo Comparator)
  Interventions: Device: Computer-controlled Local Anaesthesia (CCLA); Device: Conventional Local Anaesthesia

INTERVENTIONS:
Device: Computer-controlled Local Anaesthesia (CCLA) — The computer-controlled local anesthetic injector Calaject®, (Rønvig Dental MFG, Daugaard, Denmark), which is designed to reduce the pain of performing local anaesthesia. The principle of this device is based on the fact that the less pressure and flow of a local anaesthetic injection, the less painful will be the procedure. Each device has an installed pressure sensor as well as a three-button display that allows choosing the most appropriate program in terms of different speeds and pressure. According to the anaesthesia technique, the manufacture recommends program I for intraligamentary and palatally injections, program II for infiltration and III for alveolar nerve block techniques. Conventional carpules and needles can be used in a pen-shaped part connecting to the main unit. The administration of the anaesthetic can be achieved using a foot control pedal which is adapted to the main unit, the speed of injection is related to acoustic signals.
Device: Conventional Local Anaesthesia — Conventional dental local anaesthetic injections.

SUMMARY:
This single-blind two-arm randomized control trial (RCT) aims to evaluate the pain perception during and following administration of dental local anaesthesia using two different systems; i.e. computer-controlled (CCLA) and conventional.

DETAILED DESCRIPTION:
The administration of local anaesthesia (LA) is associated with pain, fear and anxiety. Computer-controlled LA (CCLA) aims to control the administration speed and reduce pain, fear and anxiety. This randomised control trial (RCT) aims to compare the pain perception after CCLA and conventional LA, and it uses dental students as both test and operator group versus an experienced dentist as an additional operator of the LA.

ELIGIBILITY:
Inclusion Criteria:

* Dental students at the Faculty of Medicine, University of Giessen enrolled in the course of Local Anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pain on Puncture (PoP) | Within 2 hours
  Self-reported pain intensity on puncture using visual analogue scale (0 = no pain- 10 = the worse pain)
Pain during Delivery (PdD) | Within 2 hours
  Self-reported pain intensity during delivery of the anaesthetic solution sing visual analogue scale (0 = no pain- 10 = the worse pain)

SECONDARY OUTCOMES:
Dental Anxiety (DA) | Within 2 hours
  Assessed by the Dental Anxiety Scale (DAS)- Four questions survey with five possible answers. Each answer has a score: a = 1, b = 2, c = 3, d = 4, e = 5 Total possible = 20. Anxiety rating: 9 - 12 = moderate anxiety/ 13 - 14 = high anxiety/ 15 - 20 = severe anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No